CLINICAL TRIAL: NCT01492790
Title: An Open Randomized Study Comparing Emergency Cholecystectomy First Versus Sequential Common Bile Duct Imaging/Cholecystectomy for the Management of Gallstone Migration
Brief Title: Cholecystectomy First vs Sequential Common Bile Duct Imaging + Cholecystectomy
Acronym: CCK first
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Pouya Iranmanesh, Principal Investigator, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CER 11-045 (NAC 11-012)
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Cholelithiasis; Cholecystitis
MeSH Terms: conditions — Cholelithiasis; Cholecystitis | interventions — Cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cholecystectomy first (Experimental): Patients enrolled in this arm will undergo emergency cholecystectomy first without any common bile duct imaging
  Interventions: Procedure: Emergency cholecystectomy first
- Sequential common bile duct imaging/cholecystectomy (Active Comparator): Patients enrolled in this arm will undergo common bile duct imaging and, if needed, ERCP first followed by emergency cholecystectomy
  Interventions: Procedure: Sequential common bile duct imaging/cholecystectomy

INTERVENTIONS:
Procedure: Emergency cholecystectomy first — The intervention is an emergency cholecystectomy without prior common bile duct imaging
  Arms: Cholecystectomy first
Procedure: Sequential common bile duct imaging/cholecystectomy — This intervention is a common bile duct imaging modality and, if needed, ERCP first followed in the same hospital stay by a cholecystectomy
  Arms: Sequential common bile duct imaging/cholecystectomy

SUMMARY:
The purpose of this study is to evaluate if cholecystectomy first (studied group) versus sequential common bile duct imaging/cholecystectomy (control group) result in a decrease of hospital stay, morbidity/mortality and costs in the management of patients with a suspicion of gallstone migration.

DETAILED DESCRIPTION:
Emergency cholecystectomy is nowadays an accepted surgical procedure routinely performed worldwide. The main indications include acute cholecystitis, cholangitis and gallstone migration. Abnormal liver function tests upon admission and suspicion for accompanying common bile duct (CBD) stone can delay the surgical management due to the need for further investigations and/or therapeutic maneuvers. These procedures include magnetic resonance cholangio-pancreatography (MRCP), endoscopic ultrasound (EUS) and endoscopic retrograde cholangio-pancreatography (ERCP).

While useful to detect or exclude potential CBD stones, these procedures include inherent risks, delay the surgical treatment, extend hospital stay and as a result, increase the overall medical costs. They can also potentially increase the morbidity and/or mortality by delaying emergency cholecystectomy (due to the presence of more local inflammation and adherence). Finally, more and more centers perform systematic intra-operative cholangiogram during cholecystectomies (laparoscopic or open), which allow an accurate assessment of the CBD and potentially lead to its subsequent exploration (endoscopic or surgical).

In this study, the investigators will assess the following hypotheses:

* Patients with a SUSPICION of gallstone migration (with or without associated cholecystitis) should undergo emergency cholecystectomy with intra-operative cholangiogram (IOC) first
* "Cholecystectomy first" strategy will decrease both the length of hospital stay and the morbidity/mortality by decreasing the number of unnecessary EUS, MRCP and ERCP and therefore decreasing the overall number of their complications, as well as decreasing the complications related to delayed cholecystectomy (increased adherences due to inflammation, especially in case of associated cholecystitis, which increase the risk of bleeding, CBD lesion, duodenal lesion, gastric lesion, colon lesion, gallbladder perforation and intra-abdominal gallstones spillage with potential

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a clinical diagnosis of gallstone migration, defined as right upper quadrant or epigastric abdominal pain and abnormal liver function tests (increase of at least two common hepatic parameters [AST, ALT, alkaline phosphatase, gGT and/or bilirubin], with one of them being either AST or ALT with a value at least two times higher than the norm) with a reasonable exclusion of other common differential diagnoses
* Patients will be included regardless the presence of an associated cholecystitis, defined as right upper quadrant abdominal pain, radiological signs of cholecystitis (including radiological Murphy sign and/or thickened gallbladder wall and/or free abdominal fluid around the gallbladder) and signs of infection (including fever, increased CRP or white blood cell count)
* Age ≥ 16 years

Exclusion Criteria:

* Presence of CBD stone on CT or US performed on admission (which will require ERCP exploration prior to surgery)
* Associated radiologically proven gallstone pancreatitis
* Associated cholangitis
* Medical conditions preventing surgery such as acute stroke, acute coronary syndrome, severe cardiac failure (NYHA class IV and/or respiratory failure with SpO2 < 85% with room air and/or LVEF < 35%), severe COPD with VEMS < 30 % of predicted value
* Medical conditions preventing informed consent
* Patients with contraindications to MRI (MRI-incompatible electronic devices [e.g. pacemakers], implants or prostheses, vascular clips less than 2 weeks, severe claustrophobia) and to EUS/ERCP (surgery with gastric diversion, severe cardiac dysfunction)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-06; Primary Completion 2013-02 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Hospital stay [days] | 0 - 30 days
  We will evaluate if our "new treatment" arm will have a decreased hospital stay. We do not expect patients to stay more than 30 days.

SECONDARY OUTCOMES:
Morbidity | 6 months
  We will follow-up patients until 6 months after their operation (cholecystectomy) and compare if there is any statistically significant difference between the two arms of the study in terms of morbidity.
Mortality | 6 months
  We will follow-up patients until 6 months after their operation (cholecystectomy) and compare if there is any statistically significant difference between the two arms of the study in terms of mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Pouya Iranmanesh, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

REFERENCES:
- [Derived] Iranmanesh P, Frossard JL, Mugnier-Konrad B, Morel P, Majno P, Nguyen-Tang T, Berney T, Mentha G, Toso C. Initial cholecystectomy vs sequential common duct endoscopic assessment and subsequent cholecystectomy for suspected gallstone migration: a randomized clinical trial. JAMA. 2014 Jul;312(2):137-44. doi: 10.1001/jama.2014.7587. PMID 25005650